CLINICAL TRIAL: NCT05554978
Title: Beta-blockade With Landiolol in Out-of-hospital Cardiac Arrest: a Randomized, Double-blind, Placebo-controlled, Pilot Trial
Brief Title: Beta-blockade With Landiolol in Out-of-hospital Cardiac Arrest
Acronym: Beta-Arrest
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Holzer, Principal Investigator, Professor of Emergency Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Beta Blockade Cardiac Arrest
Record Dates: First submitted 2022-04-19; First posted 2022-09-26 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; refractory; ventricular fibrillation; electrical storm; landiolol
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation | interventions — landiolol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled pilot trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: study drug preparation by a person not involved in patient recruitment and treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Landiolol (Experimental): initial dose: 20mg target dose: repeated dose (20mg) possible, max. 40mg (total)
  Interventions: Drug: Landiolol
- Placebo (Placebo Comparator): Sodium Chlorid 0,9%
  Interventions: Drug: Sodium Chloride (NaCl) 0.9%

INTERVENTIONS:
Drug: Landiolol — patient receives landiolol in addition to standard-of-care
  Other Names: Onoact; Rapibloc
  Arms: Landiolol
Drug: Sodium Chloride (NaCl) 0.9% — Placebo
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
This study investigates the efficacy of landiolol versus placebo in patients with out-of-hospital cardiac arrest (OHCA) and refractory ventricular fibrillation (electrical storm).

DETAILED DESCRIPTION:
The use of beta-blockers in OHCA patients with refractory VF could potentially reverse the unwanted beta-1-mediated effects of endogenous and exogenous epinephrine (proarrhythmic effect), which could in turn lead to a shorter time until return of spontaneous circulation (ROSC).

This is a prospective, double-blind, randomized placebo-controlled pilot trial. The investigators consider this a pilot trial, as this is the first prospective trial evaluating the use of beta-blockade in cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* OHCA , >/=18 years of age
* 3 or more shockable rhythms (VF or pVT) and last rhythm shockable

Exclusion Criteria:

* Age > 85a
* Severe head trauma or acute active bleeding
* Known allergy or insensitivity to landiolol or another beta-blocker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to sustained return of spontaneous circulation (sROSC) | Time of sROSC or termination of resuscitation efforts
  time from bolus infusion of landiolol OR placebo to sROSC

SECONDARY OUTCOMES:
rate of sustained ROSC | Time of sROSC or termination of resuscitation efforts
  number of sustained ROSC per included patients
number of shocks until sROSC | Time of sROSC or termination of resuscitation efforts
  number of shocks until sROSC per included patients
rate of temporary ROSC (any ROSC) | Time of sROSC or termination of resuscitation efforts
  number of temporary ROSC per included patients
survival to ICU admission | Time of ICU admission or termination of resuscitation efforts
  how many patients survived to ICU admission
mean/median length of stay in ICU | Time of transfer to open ward or death
  in days
mean/median length of hospital stay | Time of hospital discharge or death
  in days
survival until hospital admission | Time of hospital admission or death
  how many patients were admitted alive to the hospital
survival until hospital discharge | Time of hospital discharge or death
  how many patients survived to hospital discharge
favorable neurologic outcome at hospital discharge, day 28, month 3, 6, 12 (CPC and mRS) | at hospital discharge, day 28, month 3, 6, 12
  measured by CPC and mRS
survival at hospital discharge, day 28, month 3, 6, 12 | at hospital discharge, day 28, month 3, 6, 12
  how many patients survived to day 28, month 3, 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Holzer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
if requested, please address Georg Gelbenegger and Bernd Jilma
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after primary publication for 5 years

REFERENCES:
- See also: Department of Clinical Pharmacology — http://klpharm.meduniwien.ac.at/